CLINICAL TRIAL: NCT04496570
Title: The Role of Resolvin D1 in Maintaining Oral Health
Brief Title: Resolvin D1 Levels in Patients With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Ceren Gökmenoğlu, Principal investigator, Ordu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ordu University Dental Faculty
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Periodontitis
Keywords: gingival crevicular fluid; resolvin D1
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periodontitis patients (Active Comparator): gingival crevicular fluid and saliva collection were taken before and after nonsurgical periodontal treatment
  Interventions: Procedure: periodontal therapy
- Healthy individuals (No Intervention): gingival crevicular fluid and saliva collection were taken at baseline after oral hygiene instructions

INTERVENTIONS:
Procedure: periodontal therapy — Non surgical periodontal therapy was performed to patients with peridontitis
  Arms: Periodontitis patients

SUMMARY:
The purpose of the study was to determine the levels of Resolvin D1 (RVD1) in the gingival crevicular fluid (GCF) and saliva of the patients with periodontitis (P) and also to investigate the effects of non-surgical periodontal treatments (NSPTs) on its levels.

A total of 26 subjects (15 P, 11 healthy) were included. Clinical periodontal measurements, GCF and saliva samples were collected from each individual at baseline and 1 month after NSPTs in P group. RVD1 levels were determined by enzyme-linked immunosorbent assay (ELISA) method.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3, Grade B and generalized periodontitis patients

Exclusion Criteria:

* excessive forces;
* presence of systemic diseases
* administration of non-steroidal and anti-inflammatory drugs or antibiotic therapies within the previous 6 months
* having received non-surgical periodontal treatment within the past 6 months
* allergy or sensitivity to any drug,
* pregnancy, lactation
* current and former use of tobacco.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Biochemical parameter (resolvin D1) | Baseline and 1 month after NSPT
  The changes in levels of resolvin D1 after periodontal treatment determined by ELISA.

SECONDARY OUTCOMES:
Probing pocket depth | Baseline and 1 month after NSPT
  The changes in probing pocket depth after periodontal treatment were evaluated
Clinical attachment level (CAL) | Baseline and 1 month after NSPT
  The changes in CAL after periodontal treatment were evaluated
Plaque index (PI) | Baseline and 1 month after NSPT
  The changes in PI after periodontal treatment were evaluated
Gingival index (GI) | Baseline and 1 month after NSPT
  The changes in GI after periodontal treatment were evaluated

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)